CLINICAL TRIAL: NCT00307164
Title: A Phase II/III, Randomized, Double-Blind, Placebo-Controlled Trial of Uridine Supplementation in HIV Lipoatrophy
Brief Title: Effects of a Uridine Supplement on HIV Infected Adults With Lipoatrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5229; 10136 (Registry Identifier: DAIDS ES); ACTG A5229
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections; Lipoatrophy
Keywords: Treatment Experienced; Uridine
MeSH Terms: conditions — HIV Infections; Lipodystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- NucleomaxX (Active Comparator): Participants received NucleomaxX for 48 weeks
  Interventions: Drug: NucleomaxX
- Placebo (Placebo Comparator): Participants received NucleomaxX placebo for 48 weeks
  Interventions: Drug: NucleomaxX placebo

INTERVENTIONS:
Drug: NucleomaxX — 36 g sachet taken orally three times daily
  Arms: NucleomaxX
Drug: NucleomaxX placebo — 36 g placebo sachet taken orally three times daily
  Arms: Placebo

SUMMARY:
Lipoatrophy, the loss of body fat from particular areas of the body, is a common side effect of antiretroviral therapy (ART). The purpose of this study was to determine the effectiveness of uridine supplementation in treating HIV infected individuals on stable ART with lipoatrophy.

DETAILED DESCRIPTION:
Lipoatrophy is a distressing long-term complication of ART and is associated with decreased quality of life, an increased risk of cardiovascular disease, and nonadherence to ART. The cause of lipoatrophy in HIV-infected individuals receiving ART is not completely understood. However, past research suggests that mitochondrial toxicity in subcutaneous adipose tissue caused by thymidine analogue nucleoside analogues may be responsible for the development of lipoatrophy.

Uridine is a nucleoside that has been shown to be an effective supplement in treating individuals with mitochondrial toxicity. NucleomaxX is a food supplement that consists of mitocnol, a sugar cane extract that has a high content of nucleosides, including uridine. The purpose of this study was to evaluate the effects of uridine supplementation in the form of NucleomaxX on limb fat in HIV-infected individuals receiving stable ART containing stavudine (d4T) or zidovudine (ZDV). In addition, this study evaluated the safety and tolerability of NucleomaxX.

This study lasted for 48 weeks. Participants were randomly assigned to one of two treatment arms, stratified by d4T or ZDV use. Arm A participants received NucleomaxX for uridine, while Arm B participants received a placebo for NucleomaxX. Participants in both arms received their assigned intervention three times per day, every other day, for the duration of the study. There were 8 study visits over the 48-week study duration. Blood collection and a physical exam occurred at all study visits, and participants completed an adherence assessment at most visits. Participants underwent dual energy X-ray absorptiometry scans (DEXA) within 14 days prior to or following the screening visit and at other selected visits. Specific fasting tests for glucose and lipid levels occurred at selected visits. ART was not provided by this study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Stable ART containing zidovudine or stavudine for at least 12 consecutive weeks prior to study entry
* Cumulative ART with zidovudine or stavudine for at least 24 weeks prior to study entry
* Viral load of 5,000 copies/ml or less within 45 days prior to study entry
* Lipoatrophy in at least two of the following areas: face, arms, legs, OR buttocks
* Not planning to add to or change current vitamin supplementation
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Life expectancy of less than 12 months
* Currently enrolled in or planning to enroll in an ART interruption study
* Plans to change current ART regimen
* Liver failure at anytime prior to study entry
* Greater than Grade 2 diarrhea or vomiting within 7 days prior to study entry
* Current AIDS-defining opportunistic infection or illness. Individuals with cutaneous Kaposi's sarcoma not requiring chemotherapy are not excluded.
* Currently receiving insulin or oral hypoglycemic products for diabetes mellitus
* Systemic cancer chemotherapy or immunomodulating agents within 30 days prior to study entry
* Systemic steroids for a cumulative duration of longer than 4 weeks within the 6 months prior to study entry
* Known allergy or sensitivity to study drug or any of its components
* Severe lactose intolerance
* Current drug or alcohol abuse or dependence
* Clinically significant illness requiring systemic treatment or hospitalization
* Chronic disability or serious illness that may affect body composition
* Received an investigational drug other than NucleomaxX or uridine for lipoatrophy within 30 days prior to study entry
* Certain abnormal laboratory values
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace A. McComsey, MD, Study Chair — Division of Infectious Diseases, Case Western Reserve University; Judith A. Aberg, MD, Study Chair — New York University
Locations (30):
- United States (29):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Koch EC, Schneider J, Weis R, Penning B, Walker UA. Uridine excess does not interfere with the antiretroviral efficacy of nucleoside analogue reverse transcriptase inhibitors. Antivir Ther. 2003 Oct;8(5):485-7. No abstract available. PMID 14640397
- [Background] McComsey GA, Walker UA. Role of mitochondria in HIV lipoatrophy: insight into pathogenesis and potential therapies. Mitochondrion. 2004 Jul;4(2-3):111-8. doi: 10.1016/j.mito.2004.05.008. PMID 16120376
- [Background] Nolan D, Hammond E, Martin A, Taylor L, Herrmann S, McKinnon E, Metcalf C, Latham B, Mallal S. Mitochondrial DNA depletion and morphologic changes in adipocytes associated with nucleoside reverse transcriptase inhibitor therapy. AIDS. 2003 Jun 13;17(9):1329-38. doi: 10.1097/00002030-200306130-00007. PMID 12799554
- [Background] Walker UA, Venhoff N. Uridine in the prevention and treatment of NRTI-related mitochondrial toxicity. Antivir Ther. 2005;10 Suppl 2:M117-23. PMID 16152713
- [Result] McComsey GA, Walker UA, Budhathoki CB, Su Z, Currier JS, Kosmiski L, Naini LG, Charles S, Medvik K, Aberg JA; AIDS Clinical Trials Group A5229 Team. Uridine supplementation in the treatment of HIV lipoatrophy: results of ACTG 5229. AIDS. 2010 Oct 23;24(16):2507-15. doi: 10.1097/QAD.0b013e32833ea9bc. PMID 20827170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at AIDS Clinical Trials Units in the United States and Puerto Rico. Recruitment occurred between October 5, 2006 (date first subject was randomized) and January 7, 2008 (date last subject was randomized).
Pre-assignment Details: A total of 167 subjects were randomized, and results are reported for 165 eligible participants; two subjects never started study medication and were excluded from all analyses. The subjects were stratified by antiretroviral therapy use, stavudine (d4T) or zidovudine (AZT/ZDV).
Groups:
- NucleomaxX: Participants received NucleomaxX for uridine through week 48
- Placebo: Participants received NucleomaxX placebo through week 48
Period: Overall Study
Arm/Group | NucleomaxX | Placebo
Started | 83 | 82
Completed | 68 | 68
Not Completed | 15 | 14
Not completed — Death | 1 | 0
Not completed — Severe debilitation, unable to continue | 1 | 0
Not completed — Subject/parent not able to get to clinic | 2 | 1
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Not compliant with requirements | 4 | 4
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NucleomaxX | Placebo | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (7.78) | 48.4 (6.46) | 48.4 (7.13)
Age, Customized [Number; unit: Participants]
  30-39 Years | 9 | 10 | 19
  40-49 Years | 38 | 32 | 70
  50-59 Years | 28 | 38 | 66
  60-69 Years | 8 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 75 | 75 | 150
Race/Ethnicity, Customized [Number; unit: Participants]
  White Non-Hispanic | 50 | 52 | 102
  Black Non-Hispanic | 11 | 14 | 25
  Hispanic (Regardless of Race) | 15 | 12 | 27
  Asian, Pacific Islander | 3 | 1 | 4
  Native American, Alaskan Native | 3 | 2 | 5
  Other (More than One Race) | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 81 | 81 | 162
  Puerto Rico | 2 | 1 | 3
Antiretroviral Therapy Used (Stratification) [Number; unit: Participants]
  AZT-Containing | 63 | 63 | 126
  d4T-Containing | 20 | 19 | 39
HIV-1 RNA (copies/mL) Category [Number; unit: Participants]
  <=50 Copies | 70 | 64 | 134
  >50 Copies | 13 | 18 | 31
CD4+ Count (NucleomaxX sample size (N)=80, Placebo N=80) [Median (Inter-Quartile Range); unit: Cells/mm^3] | 506 [353 to 724] | 504 [376 to 710] | 506 [359 to 714]
Limb fat [Median (Inter-Quartile Range); unit: Grams] | 3149 [1833 to 4210] | 2995 [2082 to 4847] | 3037 [2002 to 4403]
Trunk fat [Median (Inter-Quartile Range); unit: Grams] | 8175 [5784 to 10931] | 7795 [5327 to 10825] | 8114 [5397 to 10898]
Fasting lactate (NucleomaxX N=76, Placebo N=75) [Median (Inter-Quartile Range); unit: mmol/L] | 1.3 [1.0 to 1.7] | 1.2 [0.9 to 1.5] | 1.3 [0.9 to 1.6]
Fasting glucose (NucleomaxX N=82, Placebo N=82) [Median (Inter-Quartile Range); unit: mg/dL] | 90 [84 to 98] | 87 [81 to 95] | 89 [82 to 97]
Fasting total cholesterol (NucleomaxX N=82, Placebo N=81) [Median (Inter-Quartile Range); unit: mg/dL] | 194 [163 to 216] | 190 [166 to 211] | 193 [166 to 215]
Fasting high-density lipoprotein (HDL) (NucleomaxX N=82, Placebo N=80) [Median (Inter-Quartile Range); unit: mg/dL] | 39 [33 to 49] | 37 [31 to 47] | 38 [32 to 49]
Fasting non-high-density lipoprotein (non-HDL) (NucleomaxX N=77, Placebo N=69) [Median (Inter-Quartile Range); unit: mg/dL] | 139 [123 to 168] | 145 [115 to 166] | 143 [121 to 167]
Fasting low-density lipoprotein (LDL) (NucleomaxX N=73, Placebo N=67) [Median (Inter-Quartile Range); unit: mg/dL] | 107 [88 to 132] | 110 [89 to 127] | 109 [88 to 130]
Fasting triglycerides (NucleomaxX N=82, Placebo N=81) [Median (Inter-Quartile Range); unit: mg/dL] | 161 [112 to 237] | 165 [114 to 262] | 164 [114 to 258]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 14.9 [13.7 to 15.6] | 15.0 [14.0 to 15.8] | 14.9 [13.8 to 15.7]
Leukocytes [Median (Inter-Quartile Range); unit: cells*10^3/L] | 5.6 [4.2 to 7.1] | 5.5 [4.7 to 7.0] | 5.5 [4.5 to 7.0]
Creatine kinase (NucleomaxX N=80, Placebo N=82) [Median (Inter-Quartile Range); unit: IU/L] | 125 [79 to 216] | 142 [88 to 247] | 134 [84 to 231]

OUTCOME MEASURES:

1. Primary Outcome: Change in Limb Fat (g) From Baseline
Description: Limb fat was measured at baseline and visit week 48 using dual-energy x-ray absorptiometry (DEXA), and change from baseline to week 48 (week 48 - baseline) was estimated for the treatment groups.
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with last observation carried forward (LOCF) if week 48 limb fat data was missing and post-baseline limb fat was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 75 | 69
grams | 74 [-206 to 344] | 110 [-202 to 393]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.64, Stratified Wilcoxon rank-sum test; Treatment groups were compared for change in limb fat using a two-sided stratified Wilcoxon rank-sum test (stratified by ARV used)

2. Secondary Outcome: Time to Safety Events (Signs/Symptoms or Laboratory Abnormalities)
Description: Time to safety events (grade 3 [Severe] or 4 [life-threatening] sign/symptom or laboratory-based abnormality that is at least one grade higher than baseline) from study entry
Time Frame: Through Week 48
Population: As-treated analysis with subjects stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 83 | 82
weeks | 47.1 [17.6 to 48.7] | 47.9 [34.1 to 48.7]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.17, Log Rank

3. Secondary Outcome: Number of Subjects Discontinuing Study Medication
Description: Number of eligible subjects who discontinued study medication during the study period.
Time Frame: Through Week 48
Population: Intention to treat analysis based on all subjects who started study treatment.
Measure: Number; unit: Participants
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 83 | 82
Participants | 34 | 34

4. Secondary Outcome: Change in Limb Fat From Baseline (Week 24 - Baseline)
Description: Limb fat was measured at baseline and visit week 24 using dual-energy x-ray absorptiometry (DEXA), and change from baseline to week 24 (week 24 - baseline) was estimated for the treatment groups.
Time Frame: Baseline and Week 24
Population: Intention to treat analysis with LOCF if week 24 limb fat data was missing and post-baseline before week 24 limb fat observation was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 75 | 66
grams | 54 [-117 to 315] | 7 [-202 to 238]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.25, Stratified Wilcoxon rank-sum test

5. Secondary Outcome: HIV-1 RNA Level
Time Frame: At Week 48
Population: Intention to treat analysis with all randomized subjects. Reduced sample size was due to missing data at week 48.
Measure: Number; unit: Participants
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 67 | 69
Participants
  <=50 copies/ml | 59 | 54
  >50 copies/ml | 8 | 15

6. Secondary Outcome: Change in CD4+ Count From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 CD4+ data was missing and post-baseline data was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 80 | 80
cells/mm3 | 33 [-44 to 90] | 28 [-43 to 108]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.88, Stratified Wilcoxon rank-sum test

7. Secondary Outcome: Change in Fasting Lactate From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting lactate was missing and post-baseline fasting lactate was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 67 | 62
mmol/L | 0.2 [-0.2 to 0.6] | 0.1 [-0.2 to 0.4]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.60, Stratified Wilcoxon rank-sum test

8. Secondary Outcome: Change in Fasting Glucose From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting glucose was missing and post-baseline fasting glucose was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 78 | 78
mg/dL | 2 [-6 to 9] | 4 [-5 to 11]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.13, Stratified Wilcoxon rank-sum test

9. Secondary Outcome: Change in Fasting Total Cholesterol From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting total cholesterol was missing and post-baseline fasting total cholesterol was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 77 | 75
mg/dL | 2 [-15 to 22] | -6 [-22 to 18]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.17, Stratified Wilcoxon rank-sum test

10. Secondary Outcome: Change in Fasting High-density Lipoprotein (HDL) Cholesterol From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting HDL data was missing and post-baseline fasting HDL was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 77 | 73
mg/dL | 1 [-3 to 4] | -1 [-6 to 2]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.034, Stratified Wilcoxon rank-sum test

11. Secondary Outcome: Change in Fasting Non-HDL Cholesterol From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting non-HDL data was missing and post-baseline fasting non-HDL was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF or due to associated triglyceride was >400 mg/dL. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 66 | 61
mg/dL | 2 [-13 to 18] | 2 [-18 to 17]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.76, Stratified Wilcoxon rank-sum test

12. Secondary Outcome: Change in Fasting Low-density Lipoprotein (LDL) Cholesterol From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting LDL data was missing and post-baseline fasting LDL was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 67 | 61
mg/dL | 1 [-12 to 23] | -3 [-21 to 15]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.10, Stratified Wilcoxon rank-sum test

13. Secondary Outcome: Change in Fasting Triglycerides From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 fasting triglyceride data was missing and post-baseline fasting triglyceride was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 77 | 75
mg/dL | -8 [-29 to 49] | 13 [-28 to 62]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.43, Stratified Wilcoxon rank-sum test

14. Secondary Outcome: Change in Hemoglobin From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 hemoglobin data was missing and post-baseline hemoglobin was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 83 | 81
g/dL | 0.3 [-0.5 to 0.8] | 0 [-0.8 to 0.6]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.17, Stratified Wilcoxon rank-sum test

15. Secondary Outcome: Change in Leukocytes From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 leukocyte data was missing and post-baseline leukocyte was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: cells*10^3/L
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 83 | 81
cells*10^3/L | 0.2 [-0.4 to 1.1] | 0.1 [-0.2 to 1]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.80, Stratified Wilcoxon rank-sum test

16. Secondary Outcome: Change in Creatine Kinase From Baseline (Week 48 - Baseline)
Time Frame: Baseline and Week 48
Population: Intention to treat analysis with LOCF if week 48 creatine kinase data was missing and post-baseline creatine kinase was available. Reduced sample size was due to missing baseline or missing post-baseline data for LOCF. Subjects were stratified based on ART (d4T or AZT).
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | NucleomaxX | Placebo
Number analyzed (Participants) | 79 | 81
IU/L | 1 [-39 to 45] | 5 [-31 to 68]
Statistical Analysis 1: Comparison: NucleomaxX vs Placebo; Test type: Superiority or Other; p = 0.42, Stratified Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: From treatment dispensation until off-study with variable participant follow-up time. Overall median (lower quartile, upper quartile) follow-up was 48.0 (47.7, 49.0) weeks.
Description: Grade≥2 nausea, vomiting and diarrhea and all Grade>3 signs/symptoms (S/Sx). Diagnoses per ACTG criteria for clinical events and diseases. All S/Sx or labs that led to a change in study treatment. See DAIDS Grading Severity of AEs, V1.0, Dec04, http://rcc.tech-res-intl.com
Arm/Group | NucleomaxX | Placebo
Serious Adverse Events (participants affected / at risk) | 4/83 | 2/82
Other Adverse Events (participants affected / at risk) | 75/83 | 70/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NucleomaxX (N=83) | Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NucleomaxX (N=83) | Placebo (N=82)
Diarrhoea (Gastrointestinal disorders) | 11 | 7
Nausea (Gastrointestinal disorders) | 16 | 6
Vomiting (Gastrointestinal disorders) | 7 | 3
Alanine aminotransferase increased (Investigations) | 5 | 4
Blood bilirubin increased (Investigations) | 8 | 7
Blood cholesterol (Investigations) | 5 | 4
Blood cholesterol abnormal (Investigations) | 35 | 29
Blood creatine phosphokinase increased (Investigations) | 17 | 21
Blood glucose abnormal (Investigations) | 23 | 22
Blood glucose increased (Investigations) | 6 | 3
Blood lactic acid abnormal (Investigations) | 12 | 10
Blood phosphorus decreased (Investigations) | 3 | 8
Blood triglycerides (Investigations) | 7 | 10
Low density lipoprotein abnormal (Investigations) | 28 | 16
Neuropathy peripheral (Nervous system disorders) | 26 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No